CLINICAL TRIAL: NCT05174364
Title: Epidural Versus Quadratus Lamborum Block for Postoperative Analgesia in Adult Open Nephrectomies : A Randomized Double Blind Controlled Trial
Brief Title: Epidural Versus Quadratus Lamborum Block in Adult Open Nephrectomies
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Assiut University (Other)
Responsible Party: Principal Investigator, SABastawy, M.M.B.CH & Resident Doctor at Anesthesia and Intensive Care Department, Assiut University
Other Study IDs: Open nephrectomies
Record Dates: First submitted 2021-12-14; First posted 2021-12-30 (Actual); Last update posted 2022-01-19 (Actual); Status verified 2022-01

CONDITIONS: Post Operative Analgesia

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 1 Day
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Epidural Block: Epidural block for the control group will be done before induction of general anesthesia. Patients will be positioned in the sitting position, an 18-gauge Tuohy needle will be inserted into epidural space of Th 11-12 intervertebral space under aseptic condition. In the medial approach, the site of the insertion of the needle is between the spaces created by the vertebral spinous processes. Upon locating the desired spot, lidocaine 1% must be injected into the skin and underlying tissues to decrease the discomfort with the advancement of the epidural needle
- Quadratus Lumborum Block: Bilateral QL block type 3 (anterior) for the intervention group will be performed on both sides of the patient after induction of general anesthesia. Patient will be positioned in semi-lateral decubitus and using low-frequency ultrasonography (USG) guidance attached to inferior lumbar region (Petit's triangle) that is consisted of inferior iliac crest and bordered by two muscles such as latissimus dorsi muscle in the posterior, abdominal external oblique muscle in the anterior. The USG will display the Shamrock sign, where the transverse process of vertebrae L4 role as the trunk, erector spinae muscle on the posterior side, psoas major (PM) on the anterior side, and QL muscle on the lateral side. After the visualization of QL and PM muscles, the Contiplex R needle will be directed parallel to the posterior side of the ultrasound probe until the tip of needle is confirmed in the border of QL and PM muscle

SUMMARY:
Our primary objective is to compare the effectiveness of bilateral QLB and epidural analgesia for postoperative management using VAS measured in PACU until 24 hours after surgery in patients undergoing elective open nephrectomies under GA. The secondary outcomes include: The 1st time to rescue analgesia and total amount of opioid consumption throughout the first postoperative day. hemodynamic variables. Any complications as postoperative nausea and vomiting (PONV) and sedation. The sensory block coverage & the Bromage score at 2, 6, 12, and 24 hours after anesthesia recovery and duration of urinary catheter usage. Duration of PACU stay and postoperative duration of hospitalization and Patients' satisfaction.

DETAILED DESCRIPTION:
Open surgery remains basic surgery for patients requiring radical or partial nephrectomy and is associated with a high incidence of intense immediate postoperative pain and chronic pain the months following surgery. The physiopathology of acute pain is explained as it is mediated by inflammatory cell infiltration, activation of the pain pathways in the spinal cord, and reflexive muscle spasm. All these three mechanisms of acute pain are typically ameliorated during the postoperative recovery. Regional anesthesia techniques are commonly enhanced for pain management in open nephrectomy as they decrease parenteral opioid requirements and improve patient satisfaction.

QLB has been introduced as a component of multimodal analgesia for thoracic and abdominal surgeries as:

cesarean section, hip arthroplasty, inguinal hernia repair and nephrectomies. It provides a great spread of local anesthesia which allows anesthesia from T6 - L2 and provides loss of somatic and visceral pain. The QLB was initially described by R.Blanco where the local anesthetic (LA) was injected at the anterolateral aspect of the QL muscle (type 1 QLB). Later, J.

Børglum used the posterior transmuscular approach by detecting Shamrock sign and injecting the LA at the anterior aspect of the QL (type 3 QLB). Recently, R. Blanco described another approach by injecting the LA at the posterior aspect of the QL muscle (type 2 QLB), which may be easier and safer as the LA is injected in a more superficial plane, so the risk of intra-abdominal complications and lumbar plexus injuries is less. Finally, the intramuscular QLB (type 4 QLB) was done by injecting LA directly into the QL muscle. QLBs may be particularly useful in nephrectomy as it lacks the adverse effects associated with patient controlled analgesia including nausea, vomiting, sedation, and respiratory depression, as well as side effects of patient controlled epidural analgesia such as pruritus hypotension, and urinary retention. Our hypothesis is that performing ultrasound guided QLB will be more superior or equal to epidural block in providing postoperative analgesia for patients undergoing open nephrectomy under general anesthesia

ELIGIBILITY:
Inclusion Criteria:

* Patients of American Society of Anesthesiologists (ASA) class I or II physical status.
* Age:20-60 years old.
* Patients scheduled for open nephrectomies .
* Gender: both

Exclusion Criteria:

* Patient refusal.
* Significant organ dysfunctions (e.g., cardiac, respiratory, renal, or liver disorders).
* Morbid obesity (BMI >35).
* Patient with known hypersensitivity to amide local anesthetics or morphine.
* Patient with any contraindication for intrathecal anesthesia, e.g. coagulopathy.
* Psychiatric disorders, which will make observational pain intensity assessment difficult.
* Pregnancy.
* Skin lesions or wounds at the puncture site of the proposed block .

Ages: 20 Years to 60 Years | Sex: All
Age Groups: Adult
Study Population: Any patient fulfilling the inclusion criteria participating in our study .
Sampling Method: Probability Sample
Enrollment: 62 (Estimated)
Dates: Start 2022-04-01 (Estimated); Primary Completion 2023-01-01 (Estimated); Study Completion 2023-02-01 (Estimated)

PRIMARY OUTCOMES:
compare the effectiveness of bilateral QLB and epidural analgesia | 24 hours
  postoperative pain management using visual analog scale measured in postanesthesia care unit

CONTACTS AND LOCATIONS:
Overall Officials: Kelani A. Abd El-Salam, Professor, Study Director — Assiut University

REFERENCES:
- [Background] Gupta V, Yadav SK, Dean E, Vincent P, Walid F, Al Said A. Paediatric laparoscopic orchidopexy as a novel mentorship: Training model. Afr J Paediatr Surg. 2013 Apr-Jun;10(2):117-21. doi: 10.4103/0189-6725.115035. PMID 23860059
- [Background] Bravi CA, Larcher A, Capitanio U, Mari A, Antonelli A, Artibani W, Barale M, Bertini R, Bove P, Brunocilla E, Da Pozzo L, Di Maida F, Fiori C, Gontero P, Li Marzi V, Longo N, Mirone V, Montanari E, Porpiglia F, Schiavina R, Schips L, Simeone C, Siracusano S, Terrone C, Trombetta C, Volpe A, Montorsi F, Ficarra V, Carini M, Minervini A. Perioperative Outcomes of Open, Laparoscopic, and Robotic Partial Nephrectomy: A Prospective Multicenter Observational Study (The RECORd 2 Project). Eur Urol Focus. 2021 Mar;7(2):390-396. doi: 10.1016/j.euf.2019.10.013. Epub 2019 Nov 12. PMID 31727523
- [Background] Popping DM, Zahn PK, Van Aken HK, Dasch B, Boche R, Pogatzki-Zahn EM. Effectiveness and safety of postoperative pain management: a survey of 18 925 consecutive patients between 1998 and 2006 (2nd revision): a database analysis of prospectively raised data. Br J Anaesth. 2008 Dec;101(6):832-40. doi: 10.1093/bja/aen300. Epub 2008 Oct 22. PMID 18945716
- [Background] Capdevila X, Moulard S, Plasse C, Peshaud JL, Molinari N, Dadure C, Bringuier S. Effectiveness of Epidural Analgesia, Continuous Surgical Site Analgesia, and Patient-Controlled Analgesic Morphine for Postoperative Pain Management and Hyperalgesia, Rehabilitation, and Health-Related Quality of Life After Open Nephrectomy: A Prospective, Randomized, Controlled Study. Anesth Analg. 2017 Jan;124(1):336-345. doi: 10.1213/ANE.0000000000001688. PMID 27918333
- [Background] Elsharkawy H, El-Boghdadly K, Barrington M. Quadratus Lumborum Block: Anatomical Concepts, Mechanisms, and Techniques. Anesthesiology. 2019 Feb;130(2):322-335. doi: 10.1097/ALN.0000000000002524. No abstract available. PMID 30688787
- [Background] Liu SS, Richman JM, Thirlby RC, Wu CL. Efficacy of continuous wound catheters delivering local anesthetic for postoperative analgesia: a quantitative and qualitative systematic review of randomized controlled trials. J Am Coll Surg. 2006 Dec;203(6):914-32. doi: 10.1016/j.jamcollsurg.2006.08.007. Epub 2006 Oct 25. No abstract available. PMID 17116561
- [Background] Wilkinson KM, Krige A, Brearley SG, Lane S, Scott M, Gordon AC, Carlson GL. Thoracic Epidural analgesia versus Rectus Sheath Catheters for open midline incisions in major abdominal surgery within an enhanced recovery programme (TERSC): study protocol for a randomised controlled trial. Trials. 2014 Oct 21;15:400. doi: 10.1186/1745-6215-15-400. PMID 25336055
- [Background] Dhanjal ST, Tonder S. Quadratus Lumborum Block. 2023 Aug 14. In: StatPearls [Internet]. Treasure Island (FL): StatPearls Publishing; 2025 Jan-. Available from http://www.ncbi.nlm.nih.gov/books/NBK537212/ PMID 30725897